CLINICAL TRIAL: NCT03818828
Title: A Multicenter, Open Label Phase 2 Pilot Trial of Subjects With Non-Healing Venous Leg Ulcers Treated With Standard Care Plus Cryopreserved Human Umbilical Cord (TTAX01)
Brief Title: Subjects With Non-Healing Venous Leg Ulcers Treated With Standard Care Plus Cryopreserved Human Umbilical Cord (TTAX01)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTAX01-CR002
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Venous Leg Ulcer
Keywords: venous stasis; VLU
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TTAX01 (Experimental): TTAX01 will be applied directly to the wound surface and fixed with sterile adhesive strips, plus a secondary foam dressing held in place by multi-layer compression bandaging. A single layer of the test article should cover the entire open surface of the wound. TTAX01 may overlap onto adjacent healthy tissue and must be fenestrated prior to or after fixture. The material is to be applied once every 4 weeks unless the wound shows evidence of healing, in which case product will be withheld; or, if the test article has been accidentally dislodged within 1-week post application, it may be replaced at the subsequent treatment visit.
  Interventions: Biological: TTAX01; Other: Profore Compression Therapy; Other: Cadexomer Iodine dressing

INTERVENTIONS:
Biological: TTAX01 — TTAX01 is a cryopreserved human umbilical cord product derived from donated human placental tissue following healthy, live, caesarian section, full-term births after determination of donor eligibility and placenta suitability. TTAX01 is manufactured by TissueTech Inc. utilizing a proprietary CRYOTEK® process, which devitalizes the living cells but retains the natural structural and biological characteristics relevant to this tissue. TTAX01 is aseptically processed in compliance with current Good Tissue Practices (cGTP). TTAX01 will be manufactured in various sizes, stored in a medium of Dulbecco's Modified Eagle Medium/Glycerol (1:1) containing Amphotericin B.
Other: Profore Compression Therapy — Subjects will utilize the compression system for the duration of the trial, with weekly re-applications of the compression system during study visits
Other: Cadexomer Iodine dressing — During the 2-week Screening Run-in period, subjects should be applied cadexomer iodine on the VLU.

SUMMARY:
It is hypothesized that application at 4-week intervals of the human umbilical cord tissue TTAX01 to the surface of a well debrided, nonhealing venous leg ulcer (VLU) will result in a high proportion of wounds showing complete healing within 12 weeks of initiating therapy. This open label pilot study provides a framework for a larger, controlled study. The purposes for conducting this study are to evaluate the functionality of the protocol and to obtain an estimate of product safety and efficacy when applied according to the protocol instructions, and measured according to the stated endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Age ≥ 18 years and of either sex.
* Willing to comply with protocol instructions, including allowing all study assessments.
* Have a venous leg ulcer (VLU) between the knee and ankle (at or above the malleolus), with a surface area in the range of ≥ 2.0 cm2 and ≤ 18.0 cm2 confirmed using the wound imaging and measurement device.
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence.
* Arterial supply adequacy confirmed by any one of the following: Great toe pressure ≥ 50 mm/Hg; Systolic blood pressure Ankle Brachial Index (ABI) in the range ≥ to 0.8 to ≤ 1.1; TcPO2 ≥ to 40 mmHg from the foot
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone
* Target ulcer duration ≥ 6 weeks but ≤ 104 weeks
* For diabetic subjects an HbA1C < 12.0% per the local lab report

Exclusion Criteria:

* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic).
* Deep Vein Thrombosis (DVT) that is acute, defined as the first 10 days from onset of symptoms, or any DVT for which compression bandaging is considered by the Investigator to be contraindicated.
* Clinical evidence of ulcer bed infection as described in the Study Guide.
* Documented history of osteomyelitis at the target wound location within 6 months preceding the Screening Visit.
* Refusal of or inability to tolerate compression therapy.
* The subject is pregnant
* The subject is a nursing mother
* The subject is a woman of child-bearing potential who is unwilling to avoid pregnancy or use an appropriate form of birth control (adequate birth control methods are defined as: topical, oral, implantable, or injectable contraceptives; spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or surgical sterilization of partner).
* Therapy of the target ulcer with other birth tissue products, autologous skin graft, Apligraf®, or Dermagraft® within 30 days preceding the Screening Visit.
* Therapy of the target ulcer with topical growth factors within 1 week preceding the Screening Visit.
* Current therapy with systemic antibiotics.
* Current systemic therapy with cytotoxic drugs.
* Current therapy with chronic (> 10 days) oral corticosteroids.
* Current therapy with TNF alpha inhibitors other than Trental® (pentoxifylline).
* History of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers).
* The subject has had previous use of NEOX® CORD 1K®, CLARIX® CORD 1K®, or TTAX01 applied to the index ulcer
* The subject has an allergy to Amphotericin B or glycerol
* The subject has an allergy to primary or secondary dressing materials used in this trial
* Per Investigator's discretion the subject is not appropriate for inclusion in the trial, e.g., undergoing surgical treatments or the subject currently has sepsis, i.e., life-threatening organ dysfunction caused by a dysregulated host response to infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Complete wound healing | 12-weeks
  Proportion of subjects who achieve complete wound closure over the 12-week treatment period from baseline with a 4 week followup to confirm wound healing.

SECONDARY OUTCOMES:
Time to complete wound healing | up to 12 weeks
  Time, in days, from baseline to initial observation of closure, in cases where healing is later confirmed.
Complete wound healing | up to 12 weeks
  Proportion of subjects with complete wound closure at each of the 12 treatment weeks from baseline
Changes in pain using the numeric rating scale | up to 12 weeks
  Change from baseline in pain level as reported using a numeric rating scale for the target ulcer and the affected leg, separately. Subjects will be asked to rate the level of pain they experience on a scale from 0 to 10, with 0 representing "no pain" and 10 representing "the worst possible pain".

OTHER OUTCOMES:
Sheffield Preference-based Venous Ulcer questionnaire (SPVU-5D) quality of life questionnaire | up to 17 weeks
  The SPVU-5D is a condition-specific preference-based measure of health-related quality of life for use in the assessment of the impact of venous ulceration. It has five dimensions encompassing physical, psychological and social aspects. The dimensions have between three and five levels. The measure was developed from the bottom-up and incorporates items generated from patients. The measure has been shown to have good practicality and validity. Preference-weights and a scoring algorithm were produced based on valuations from the UK population.

CONTACTS AND LOCATIONS:
Overall Officials: Scheffer Tseng, MD, PhD, Study Chair — Chief Technology Officer
Locations (6):
- United States (6):
  - ILD Consulting, Inc., Carlsbad, California
  - UCLA Olive View, Sylmar, California
  - Rosalind Franklin University, North Chicago, Illinois
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - St Luke's-Roosevelt Hospital Center, New York, New York
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No